CLINICAL TRIAL: NCT06260332
Title: Move Toward Recovery: A Physical Activity Intervention to Reduce Persistent Pain Following Breast Surgery for Cancer in Young, Hispanic Women
Brief Title: Physical Activity Intervention for the Improvement of Pain in Young, Hispanic Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INST UNM 2302; 23-293 (Other: UNM HSC IRB)
Record Dates: First submitted 2024-01-23; First posted 2024-02-15 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Fitbit) (Experimental): Patients wear a Fitbit and use the Fitbit application to monitor their physical activity daily in weeks 2-12 with the goal of increasing their number of steps per day and their number of active hours per day. Starting at week 2, patients also receive educational materials and attend 6 calls over 20-60 minutes each with their health coach in weeks 2, 3, 5, 7, 9, and 11.
  Interventions: Behavioral: Supportive Care (Fitbit)

INTERVENTIONS:
Behavioral: Supportive Care (Fitbit) — Wear Fitbit, Use Fitbit application, Receive educational materials, attend coaching calls, Ancillary studies
  Other Names: Medical Device Usage and Evaluation; Internet-Based Intervention; Educational Activity; Counseling; Survey Administration

SUMMARY:
This clinical trial tests whether increased activity throughout the day can improve the chronic pain and associated symptoms that breast cancer survivors may experience after surgery. Staying active is a key factor of one's physical, mental, and social health and well-being. Moving more could also reduce pain and associated stress, anxiety, or depression. Using a fitness tracker may help patients to move around more, whether or not they choose to exercise. Information gathered from this study may help researchers learn how the use of a Fitbit tracker with health coaching may improve physical activity and reduce pain in young, Hispanic breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of a physical activity intervention in young, Hispanic women with chronic post-operative pain after breast surgery for invasive breast cancer, termed post breast surgery pain syndrome (PBSPS) for this study.

SECONDARY OBJECTIVES:

I. To assess the preliminary efficacy of a physical activity intervention in decreasing pain in young, Hispanic women with PBSPS.

II. To assess the preliminary efficacy of the physical activity intervention in increasing physical activity and improving health-related quality of life (hrQOL).

OUTLINE:

Patients wear a Fitbit and use the Fitbit application to monitor their physical activity daily in weeks 2-12 with the goal of increasing their number of steps per day and their number of active hours per day. Starting at week 2, patients also receive educational materials and attend 6 calls over 20-60 minutes each with their health coach in weeks 2, 3, 5, 7, 9, and 11.

ELIGIBILITY:
Inclusion Criteria:

* Women who have completed surgery for invasive breast cancer >= 6 months prior to enrollment
* Any breast surgery (lumpectomy or mastectomy)
* Baseline low to moderate activity level (exercise less than 120 minutes a week)
* PBSPS defined as pain in the area of breast surgery of at least moderate intensity (>= 4 on a scale of 1-10), located in the ipsilateral beast/chest wall, axilla or arm, lasting at least 6 months, and occurring at least 50% of the time
* Self-identified as Hispanic/Latinx
* Age, >= 18 and =< 60 years
* Endocrine therapy and ovarian suppression is allowed

Exclusion Criteria:

* Metastatic or locally recurrent disease with no option for curative intent treatment
* Meeting or exceeding physical activity guidelines (> 150 minutes per week of moderate-intensity exercise)
* Unable to speak, read, and understand English or Spanish
* Severe impairments (in seeing or hearing) or pre-existing medical limitations for engaging in daily physical activity. This is defined as the ability to walk 3 blocks without stopping to rest and without using an assistive device
* Unwilling to use a study provided smartphone (if do not already own one) and wear activity trackers/monitors
* Adults not able to consent are excluded from participation
* Based on the age criteria (18 years and older), individuals who are not yet adults (infants, children, teenagers) may not participate in this study due to the same age criteria above
* Pregnant women
* Prisoners may not participate in this study as this is a study of free-living individuals

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 25 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate (Feasibility) | Up to 1 year
  This study will be considered feasible with the recruitment of 25 breast cancer patients.
Retention rate (Feasibility) | Up to 12 weeks
  This study will be considered feasible if 80% of patients complete all pre and post assessments.
Adherence rate (Feasibility) | Up to 12 weeks
  This study will be considered feasible if participants complete at least 4 of 5 health coaching sessions (80%).
Incidence of adverse events | Up to 12 weeks
  Safety will be tracked by the study team.

SECONDARY OUTCOMES:
Change in chronic post-surgical pain | At 13 weeks
  Reducing chronic post-surgical pain will be measured using the Defense and Veterans Pain Rating Scale. Will also be assessed by Bodily Threat Monitoring Scale and pain self-efficacy questionnaire. Will summarize change scores with means and standard deviations, or medians and interquartile ranges, and obtain 95% confidence intervals. Will perform one-sided paired t-tests, or Wilcoxon signed rank tests.
Change in physical activity | At 13 weeks
  Increasing physical activity will be measured using accelerometry data using the activePAL activity monitor. Will summarize change scores with means and standard deviations, or medians and interquartile ranges, and obtain 95% confidence intervals. Will perform one-sided paired t-tests, or Wilcoxon signed rank tests.
Change in health-related quality of life (hrQOL) | At 13 weeks
  Improvement in hrQOL will be measured using Patient-Reported Outcomes Measurement Information System surveys. Will summarize change scores with means and standard deviations, or medians and interquartile ranges, and obtain 95% confidence intervals. Will perform one-sided paired t-tests, or Wilcoxon signed rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jacklyn M Nemunaitis, MD, Principal Investigator — New Mexico Cancer Research Alliance; Cindy K Blair, Ph.D., Principal Investigator — New Mexico Cancer Research Alliance
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH. (n.d.). Cancer of the breast (female) - cancer stat facts. SEER. Retrieved January 22, 2023 — https://seer.cancer.gov/statfacts/html/breast.html
- See also: PROMIS: Patient-Reported Outcomes Measurement Information System — http://www.healthmeasures.net/explore-measurement-systems/promis/intro-to-promis